CLINICAL TRIAL: NCT04386122
Title: An in Vivo Bioequivalence Study of FABALOFEN 60 (Loxoprofen Sodium 60mg/Tablet) of Pharbaco Central Pharmaceutical J.S.C No.I With JAPROLOX® TABLETS (Loxoprofen Sodium 60mg/Tablet) of Daiichi Sankyo Propharma Co., Ltd
Brief Title: An in Vivo Bioequivalence Study of 2 Loxoprofen Sodium Products in Vietnamese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre of Clinical Pharmacology, Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCP2018-BE.07
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Bioequivalence
MeSH Terms: interventions — loxoprofen; Tablets

STUDY DESIGN:
Intervention Model Description: A randomized, single-dose, 2-sequence, 2-period, 2-treatment crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FABALOFEN 60 (Experimental): Subjects will receive a single dose of 1 FABALOFEN 60 tablet under fed condition
  Interventions: Drug: FABALOFEN 60
- JAPROLOX TABLET (Active Comparator): Subjects will receive a single dose of 1 JAPROLOX® TABLETS tablet under fed condition
  Interventions: Drug: JAPROLOX TABLET

INTERVENTIONS:
Drug: FABALOFEN 60 — Dosage: Single dose of one tablet of test product in each period. Administration: 30 minutes before administration, subjects will receive a test meal (high-fat and high-calorie) and finish this meal in 30 minutes or less. Take 1 tablet of test product with 240 mL of water. Lying position or strenuous activities are not allowed within 2 hours post dose
  Other Names: Loxoprofen sodium 60mg/tablet
  Arms: FABALOFEN 60
Drug: JAPROLOX TABLET — Dosage: Single dose of one tablet of reference product in each period. Administration: 30 minutes before administration, subjects will receive a test meal (high-fat and high-calorie) and finish this meal in 30 minutes or less. Take 1 tablet of reference product with 240 mL of water. Lying position or strenuous activities are not allowed within 2 hours post dose
  Other Names: Loxoprofen sodium 60mg/tablet
  Arms: JAPROLOX TABLET

SUMMARY:
This study aims to investigate whether FABALOFEN 60 is bioequivalent to JAPROLOX® TABLETS after a single oral administration of each loxoprofen formulation in healthy subjects by assessing of pharmacokinetic properties including AUC, Tmax and Cmax and to evaluate the safety of test drug FABALOFEN 60 and reference drug JAPROLOX® TABLETS during drug administration.

DETAILED DESCRIPTION:
This study is a randomized, single-dose, 2-sequence, 2-period, 2-treatment crossover study in 24 fed healthy subjects with an at-least-6-day washout period. The drug level in serum is detected by High-performance Liquid Chromatography (HPLC) to determine Cmax, AUC0-t and Tmax. Safety are evaluated during drug administration, blood sampling time, washout period and 1 week after the end of blood sampling for any adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males.
* 18 to 55 years old.
* BMI in the range of 18 - 27 kg/m2, according to 1983 Metropolitan Index for adults.
* No present or history of hypertension, diabetes, respiratory or digestive problems, hepatic or renal deficiency, genetic problems nor tuberculosis (all inclusive).
* Laboratory results (hematological, biological) within normal range; negative HIV-test and HbsAg.
* No abnormalities on ECG.
* Willing to participate in the study.

Exclusion Criteria:

* Legal incompetency.
* Drug, alcohol or tobacco abuse.
* Allergic history to loxoprofen or any other excipients of the study products, or heparin.
* Abnormalities in cardiovascular, digestive, immunity, hematological, endocrine, neurological or psychiatric system determined by clinical physicians.
* Suspected positive HIV-test or HbsAg by quick test or electrochemiluminescence Immunoassay (ECLIA) or enzyme-linked immunosorbent assay (ELISA).
* Any illness determined by clinical physicians within 2 weeks prior to the first dosing.
* Use of any over-the-counter drug within 1 week or prescription drug within 2 weeks prior to the first dosing.
* Donation or loss of more than 450 ml of blood within 28 days prior to the first dosing.
* History of dysphagia or digestive diseases affecting drug absorption.
* History of difficulty in accessibility of veins in arms.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-05-17 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Up to 8 hours post-administration
  Area under the plasma concentration curve from time 0 to the last measured (AUC0-t). Analyzing AUC with ANOVA test to evaluate the 90% confidence interval for the ratio (Test/Reference) of the population mean with a logarithmic transformation prior to analysis with acceptance interval of 0.80 - 1.25.
Cmax | Up to 8 hours post-administration
  Maximum plasma concentration. Analyzing Cmax with ANOVA test to evaluate the 90% confidence interval for the ratio (Test/Reference) of the population means with a logarithmic transformation prior to analysis with acceptance interval of 0.80 - 1.25.
Tmax | Up to 8 hours post-administration
  Time until Cmax is reached. Tmax is analyzed with Wilcoxon non-parametric test

SECONDARY OUTCOMES:
Adverse Events | Up to approximately 14 days
  The number and type of adverse events will be reported from first drug administration (period 1) till 1 week after the second drug administration (period 2), including 6 days of washout period (total time is approximately 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh P Nguyen, MD, Principal Investigator — Centre of Clinical Pharmacology, Hanoi Medical University
Locations (1):
- Centre of Clinical Pharmacology, Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No